CLINICAL TRIAL: NCT01395264
Title: Saccadometry in Primary Headache Syndromes
Status: Terminated | Type: Observational
Why Stopped: Lack of available clinical time to complete
Sponsor: Tim Young (Other)
Responsible Party: Sponsor-Investigator, Tim Young, Doctor, University College London Hospitals
Organization: University College London Hospitals (Other)
Other Study IDs: 10/0366
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Migraine; Cluster Headache; Control; Menstrual Migraine
MeSH Terms: conditions — Migraine Disorders; Cluster Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Episodic Migraine.
- menstrual migraine
- Cluster Headache patients
- control (non-headache group)

SUMMARY:
Migraine is one of the commonest neurological disorders, affecting up to 12% of the general population, but remains relatively under-diagnosed and under-treated. Migraine has a wide socioeconomic impact and brings a large economic burden; estimates suggest that disability due to migraine costs > €27 billion per annum across Europe. Despite its prevalence and impact, migraine pathophysiology is poorly understood. A wider understanding of the functional changes in this disorder would be beneficial to both diagnosis and treatment.

Saccades are the rapid eye movements we make when moving the eyes to a new object in our visual field. Reaction time studies have been used to investigate Huntington's disease and Parkinson's disease with great success. These use saccadic tasks (monitoring eye movements). Even at rest we make approximately three saccades per second, so a lot of data can quickly be gathered with non-invasive testing. We hope to understand more of the underlying mechanisms of migraine by studying reaction time in migraine patients.

Our previous pilot study, with less stringent inclusion and exclusion criteria, looked at fewer patients (32 migraineurs and 32 controls), and found that migraineurs showed significantly different saccadic patterns to non-migraineurs.

This study firstly seeks to corroborate the saccadometric findings of our earlier pilot study in a group of migraineurs, and secondly to explore the specificity of these findings in migraine by also studying patients with another primary headache syndrome, namely cluster headache.

Migraine is known to be a dynamic disorder, with previous studies showing longitudinal changes in the migraine brain. To explore this further we hope to record longitudinally (Every day for 21 days) in a small subset of migraineurs to identify potential longitudinal changes in saccadic reaction time. Because of the portability of the equipment this could be done in the subjects own home if they preferred.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and aged between 18 and 60 years in good general health apart from suffering from headaches (test group).
2. Migraine and cluster headache will be diagnosed according to ICHD-II diagnostic criteria (6).
3. Migraineurs must suffer at least two migraine attacks per year and no more than 5 attacks per month.

   -

Exclusion Criteria:

1. Any other neurological disorder such as stroke, multiple sclerosis, epilepsy, concussion within the past year, psychiatric disorders, visual disorders.
2. Use of migraine prophylactic medication in the last month or acute migraine therapy in the 3 days prior to testing.
3. Patients on any medication to treat depression in their case
4. Headache during testing or within 3 days before and after testing.

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: From hospital Headache clinics (secondary and tertiary)
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-08; Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
To see if Saccadometry results differ between controls and migraine subjects | By May 2019

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Neurology Department, Whittington Hospital, London
  - The National Hospital for Neurology and Neurosurgery, London WC1N 3BG, and The John Radcliffe hospital, Oxford, The Whittington Hospital N19 5NF London, London